CLINICAL TRIAL: NCT05168280
Title: Intraoperative Infusion of Dexmedetomidine for Prevention of Postoperative Delirium in Elderly Patients Undergoing Craniotomy: a Randomized Clinical Trial
Brief Title: Intraoperative Infusion of Dexmedetomidine for Prevention of Postoperative Delirium in Elderly Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Tiantan Hospital (Other)
Responsible Party: Principal Investigator, Yuming Peng, Deputy chief of Department of Anesthesiology, Beijing Tiantan Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2021-12-05
Record Dates: First submitted 2021-12-13; First posted 2021-12-23 (Actual); Last update posted 2025-03-03 (Actual); Status verified 2025-02

CONDITIONS: Dexmedetomidine; Postoperative Delirium
MeSH Terms: conditions — Emergence Delirium | interventions — Dexmedetomidine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DEX group (Active Comparator): The DEX group patients will be received dexmedetomidine intraoperatively.
  Interventions: Drug: Dexmedetomidine
- Placebo group (Placebo Comparator): The placebo group patients will be received 0.9% saline intraoperatively.
  Interventions: Drug: 0.9% saline

INTERVENTIONS:
Drug: Dexmedetomidine — The 200ug dexmedetomidine will be diluted into a 50ml syringe and administered with 0.4ug/kg/h intraoperatively.
  Arms: DEX group
Drug: 0.9% saline — The 0.9% saline is administered with the same volume at the same speed as the other group.
  Arms: Placebo group

SUMMARY:
Postoperative delirium (POD) is a common surgical complication. The incidence is 10% to 22% in neurological procedures, and advanced age is a risk factor for neurological procedures. Many studies have shown that dexmedetomidine(DEX) may reduce the incidence of delirium in non-cardiac surgery patients and elderly patients. However, there are few studies focus on the effect of DEX on POD in elderly patients undergoing neurosurgery. The purpose of this study was to investigate the effect of DEX on POD in in elderly patients undergoing craniotomy.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing selective craniotomy.
* Age ≥65 years.
* Obtain written informed consent.

Exclusion Criteria:

* Operation time less than 2 hours.
* Refusal to provide written informed consent.
* Cognitive impairment before surgery(mini-mental state examination, MMSE ≤ 26 or Montreal Cognitive Assessment, MoCA≤22).
* Allergic to the study drug.
* Body mass index ≤18 or ≥ 30 kg/m2.
* History of psychotropic drugs, anticholinergic drugs, antihistamine drug and dopaminergic drugs.
* History of traumatic brain injury or neurosurgery.
* Severe bradycardia (heart rate less than 40 beats per minute), sick sinus syndrome or second-to-third degree atrioventricular block.
* Severe liver dysfunction (Child-Pugh grade C) or renal failure (requiring kidney replacement therapy).
* The functional neurosurgery.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 420 (Estimated)
Dates: Start 2022-07-18 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
The incidence of postoperative delirium | postoperative 5 day
  Postoperative delirium is assessed by the combination of the Richmond Anxiety Scale (RASS) and the Confusion assessment method for intensive care unit (CAM-ICU) or the 3-minute diagnostic interview for CAM (3D-CAM) as applicable.
  Delirium consists of four main characteristics: acute onset of a change in mental status or a fluctuating level of consciousness, inattention, disorganized thinking and an altered level of consciousness. The patient was diagnosed as delirious if both the first and second features were present, and either the third or fourth was present.
  In the ICU, the delirium assessment was performed in two steps. The arousal level was first assessed by RASS. If the patient was not responsive to verbal stimuli (i.e. RASS score ≤-4), the remaining delirium assessment was aborted, and the patient was recorded as comatose. When the RASS score was greater than or equal to 3, delirium was evaluated using the CAM-ICU. Patients in general ward were evaluated by 3D-CAM.

SECONDARY OUTCOMES:
Pain severity score | postoperative 5 day
  The degree of surgical incision pain will be assessed at rest and on movement by Numerical Rating Scale (NRS). NRS ranges from 0 to 10, with the highest score indicating the worst pain.
The quality of recovery | postoperative 1 day
  The quality of recovery will be assessed with 15-item quality of recovery questionnaire (QoR-15). The QoR-15 measures cognitive function, physical activity, language and mood on a 150-point scale, with higher scores indicating better quality of recovery.
The quality of sleep | postoperative 3 day
  The quality of sleep will be assessed by the Richards Campbell sleep questionnaire (RCSQ).RCSQ is mainly used to evaluate the sleep quality of the previous night. The scale comprises five items: sleep depth, sleep latency, wake up times, relapse to sleep and overall sleep quality.The total score of the scale is the average of 5 items, and the lower the score, the better the sleep quality.
Cognitive function | 1 day before surgery and 5 days after surgery
  Cognitive function will be assessed 1 day before surgery and 5 days after surgery using MMSE scale and Montreal Cognitive Assessment (MoCA) scale. MMSE includes seven items: time orientation, place orientation, immediate memory, attention and calculation, delayed memory, language and visual space.A total of 30 questions will be asked, 1 point for each correct answer, 0 point for a wrong answer or unknown answer and the total score range from 0 to 30. MoCA scale was widely identified that MoCA was superior to MMSE in the detection of mild cognitive impairment. Furthermore, the MoCA showed differences in cognitive profile even in those performing in the normal range on the MMSE and would appear to be a useful brief tool to assess cognition in those with mild cognitive impairment.
Psychological health state | 1 day before surgery and postoperative 5 day
  Psychological health state will be assessed by Generalized Anxiety Disorder-7 (GAD-7) and Patient Health Questionnaire-9 (PHQ-9).There are 7 and 9 items to screen anxiety and depression, respectively. The point of each item is 3. The total points >4 will be regarded as anxiety and depression.
The intraoperative data | The surgery day
  Intraoperative data include total dose of anesthetics, bispectral index scale value, and cardiovascular adverse events will be recorded and classified as hypotension (systolic blood pressure<95mmHg, or lower than 30% baseline), hypertension (systolic blood pressure ≥180 mmHg, or higher than 30% baseline), bradycardia (heart rate <40 beats /min), tachycardia (heart rate ≥ 100 beats /min) or hypoxemia (pulse oxygen saturation<90%).
Length of stay in ICU and hospital, hospitalization costs, and non-delirium complications. | postoperative 5 day
  Non-delirium complications include cardiac arrest, infection of the incision, sepsis, intracranial hematoma, severe intracranial edema (base on brain images), stroke, myocardial infarction, pulmonary infection and embolism.
30-day all-cause mortality | postoperative 30 day
  Postoperative 30-day all-cause mortality.
The physiological status | 1 day before surgery
  The physiological status of the patients will be assessed by Short-Form Mini-nutrition assessment (MNA-SF) and FRAIL scale.
Electroencephalogram changes | The surgery day
  Electroencephalogram will be used to record the brain activity.
Regional cerebral oxygen saturation changes | The surgery day
  Regional cerebral oxygen saturation will be monitored with near-infrared spectroscopy.

CONTACTS AND LOCATIONS:
Overall Officials: Yuming Peng, MD,Ph.D, Principal Investigator — Beijing Tian Tan Hospital
Locations (1):
- Beijing Tian Tan Hospital, Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
Study protocol and de-identified individual participant data could be shared after 1 year after publication with the permission of principle investigator for reasonable usage.
Supporting Information: Study Protocol
Time Frame: The data could be shared after 1 year after publication with the permission of principle investigator. The duration of the data sharing will be determined by principle investigator after publication.
Access Criteria: Study protocol and de-identified individual participant data could be shared after 1 year after publication with the permission of principle investigator. Please email principle investigator if researchers wish to have the data.

REFERENCES:
- [Derived] Cui Q, Ma T, Liu M, Shen Z, Li S, Zeng M, Liu X, Zhang L, Peng Y. Intraoperative infusion of dexmedetomidine for prevention of postoperative delirium in elderly patients undergoing craniotomy: a protocol of randomised clinical trial. BMJ Open. 2023 Jan 23;13(1):e063976. doi: 10.1136/bmjopen-2022-063976. PMID 36690404